CLINICAL TRIAL: NCT00955370
Title: The Experience of Uncertainty in Parents of Children With an Undiagnosed Medical Condition
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909206; 09-HG-N206
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-10

CONDITIONS: Multiple Abnormalities
Keywords: Uncertainty; Undiagnosed; Rare Diseases; Parents; Multiple Abnormalities
MeSH Terms: conditions — Abnormalities, Multiple; Rare Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

* Rare and undiagnosed conditions are often chronic and disabling, with symptoms affecting different organ systems at various levels of severity. Perhaps the most challenging feature of an undiagnosed medical condition that has lasted 2 or more years is its characteristic uncertainty. In the absence of a diagnosis, health care professionals can provide only limited treatment and prognostic information.
* In the case of a child with an undiagnosed condition, the uncertainty that accompanies what is often a chronic, debilitating medical condition and an undefined prognosis may have physical, psychological, social, and spiritual implications for the entire family. Research suggests that parents of a child with an undiagnosed medical condition may be at significantly increased risk of anxiety, depression, poor health, and overall lower quality of life.
* It is not well understood how individuals cope with and adapt to chronic uncertainty, and the factors that influence this process. To design future interventions, descriptive studies are needed to reveal predictors that can be manipulated to improve outcomes.

Objectives:

* To examine whether perceptions of uncertainty, and perceived personal control, are associated with coping and adaptation.
* To examine how the length of time elapsed since child was identified as sick and perceptions of uncertainty affect coping and adaptation.
* To assess how perceptions of uncertainty, time elapsed since child became sick, optimism, and perceived personal control affect coping and adaptation.

Eligibility:

* Parents (older than 18 years of age) of children who have an undiagnosed medical condition.
* Participants must have a working e-mail address or fixed postal address.

Design:

* Parents will be recruited from Web-based support networks for parents of undiagnosed children through Web site postings, electronic mailing lists, and printed newsletter postings.
* Participants will be asked to complete a questionnaire about their experiences in living with a child who has an undiagnosed but chronic medical condition. The main outcome variable is adaptation to living with one's child's undiagnosed medical condition.
* Participants have the option to complete an online or paper version of the questionnaire. The questionnaire should take between 20 and 30 minutes to complete.
* No medical treatments are specifically offered as a part of this study.

DETAILED DESCRIPTION:
This study aims to understand the impact on parents of having a child with an undiagnosed medical condition and the factors that contribute to their adaptation. Rare and undiagnosed conditions are often chronic and disabling, with symptoms affecting different organ systems at various levels of severity. Perhaps the most challenging feature of an undiagnosed medical condition that has lasted two or more years, however, is its characteristic uncertainty. In the absence of a diagnosis, health care professionals can provide only limited treatment and prognostic information. It is not well understood how individuals cope with and adapt to chronic uncertainty, and the factors that influence this process. To design future interventions, descriptive studies are needed to reveal predictors that can be manipulated to improve outcomes. In this study, Lazarus and Folkman's Transactional Model of Stress and Coping provides a framework to examine coping and adaptation in the parents of children who have had a chronic, undiagnosed medical condition for two or more years. A cross-sectional research design using a mixed methods survey will be used to examine the relationships among appraisals (perceptions of uncertainty and perceived personal control), time elapsed since parents first realized their child was sick, coping and adaptation. Parents will be recruited from web-based support networks for parents of undiagnosed children via website postings, email listservs and printed newsletter postings. Participants will have the option to complete an online or paper version of the questionnaire. The main outcome variable is adaptation to living with one's child's undiagnosed medical condition.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Men and women 18 years or older
* Biological or adoptive parent
* At least one child of participants has a medical problem or problems that have remained undiagnosed for > 2 years
* The child with an undiagnosed medical problem must reside with the parent
* Read and write in English

EXCLUSION CRITERIA:

-One parent/household may participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-08-04; Study Completion 2012-04-10

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Guillem P, Cans C, Robert-Gnansia E, Ayme S, Jouk PS. Rare diseases in disabled children: an epidemiological survey. Arch Dis Child. 2008 Feb;93(2):115-8. doi: 10.1136/adc.2006.104455. Epub 2007 Oct 17. PMID 17942587
- [Background] Lenhard W, Breitenbach E, Ebert H, Schindelhauer-Deutscher HJ, Henn W. Psychological benefit of diagnostic certainty for mothers of children with disabilities: lessons from Down syndrome. Am J Med Genet A. 2005 Mar 1;133A(2):170-5. doi: 10.1002/ajmg.a.30571. PMID 15666306
- [Background] Rosenthal ET, Biesecker LG, Biesecker BB. Parental attitudes toward a diagnosis in children with unidentified multiple congenital anomaly syndromes. Am J Med Genet. 2001 Oct 1;103(2):106-14. doi: 10.1002/ajmg.1527. PMID 11568915